CLINICAL TRIAL: NCT04490109
Title: A Phase II, Randomized, Double-Blind, Vehicle Controlled Study of the Efficacy, Safety, and Tolerability of B244 Topical Spray for the Treatment of Pruritus in Adults With a History of Atopic Dermatitis
Brief Title: B244 Topical Spray for the Treatment of Pruritus in Adults With a History of Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AOBiome LLC (Industry)
Collaborators: bioRASI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRB244-01
Record Dates: First submitted 2020-07-16; First posted 2020-07-28 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Atopic Dermatitis; Pruritus
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, randomized, vehicle-controlled, randomized in a 1:1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- B244 Suspension O.D. 5.0 (Experimental): One arm of 192 Subjects will be receiving a dose of B244 O.D. 5.0 suspension
  Interventions: Biological: B244
- B244 Suspension O.D. 20.0 (Experimental): Second arm of 192 subjects will receive a dose of B244 O.D. 20.0 suspension
  Interventions: Biological: B244
- Placebo (Placebo Comparator): Third arm of 192 subjects will receive a vehicle dosing.
  Interventions: Biological: Vehicle

INTERVENTIONS:
Biological: B244 — B244 suspension
  Arms: B244 Suspension O.D. 20.0; B244 Suspension O.D. 5.0
Biological: Vehicle — Vehicle suspension
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, vehicle-controlled study to assess the efficacy, safety, and tolerability of 2 doses of B244 for the treatment of pruritus in adults with a history of atopic dermatitis. Subjects who meet the study entry criteria will be randomized in a 1:1:1 ratio to receive twice daily topical doses of B244 O.D. 5.0, B244 O.D. 20.0, or vehicle (placebo) for 4 weeks.

DETAILED DESCRIPTION:
This is a Prospective, Vehicle Controlled, Double-Blind, Multicenter, Randomized Phase II Trial, comparing the effect of twice daily B244 applications for 4 weeks vs vehicle applications on treatment of mild to moderate pruritus associated with atopic dermatitis.

* Approximately 576 subjects may be enrolled.
* The total duration of the study will be approximately 11 weeks. Participants will report for a Screening visit and if all inclusion/exclusion criteria are met, subjects will go through a two-week washout phase before reporting for a Baseline visit.
* After screening and baseline, participants will be randomized to one of two doses of B244 or vehicle application for 4 weeks.
* Randomization will be 1:1:1 so that an equal number of patients will be treated in each Arm of the study.
* All B244 randomized subjects will be treated at the dose of O.D. 5.0 or O.D. 20.0
* Subjects must be willing and able to complete diary within a consistent time frame on a daily basis and to comply with restrictions on allowable therapies for the duration of the study.
* All subjects will attend a screening visit not more than 21 days prior to Baseline (Day 0).
* Subjects will be required to return to the clinic at Baseline, Day 14 (Week 2) and Day 28 (Week 4) visits. All subjects will be asked to attend a Week 8 follow-up visit 4 weeks (28 (±3) days) after the last dose of study medication.
* Subjects will apply a total of 10 pumps of IP per application across all affected areas twice-a-day (i.e. 10 pumps in the morning and 10 pumps again at night) for 4 weeks.
* Safety evaluations will consist of review of participant's medical history at screening and on-going assessment of adverse events reported throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 to 65 years of age.
2. Pruritus of at least 4 weeks duration prior to the initial Screening visit and during the 2 week washout period.

   a. Subjects using stable doses of oral H1 antihistamines at the initial Screening visit must be willing to continue these at the same doses and frequencies throughout the study inclusive of the follow-up period.
3. Worst Itch Numeric Rating Scale (WI-NRS) score ≥ 7 in the 24-hour period prior to the initial Screening as well as Baseline visits.
4. Average weekly WI-NRS score ≥6 for each week of the washout period, as recorded in the eDiary.
5. A history of atopic dermatitis for greater than 12 months consistent with a diagnosis of atopic dermatitis, as defined by the 2014 American Academy of Dermatology (AAD) Guidelines of Care for the Management of Atopic Dermatitis.

   1. Subjects using bland emollients at the initial Screening visit will be allowed to continue to use their emollient of choice at the same dose and frequency throughout the study.
   2. Subjects using low- to mid-potency topical corticosteroids at the initial Screening visit will be allowed to use their topical corticosteroid of choice at the same dose and frequency no more than 7 days per month throughout the study as rescue medication.
6. A minimum of 10% and not more than 40% of the subjects' BSA affected by atopic dermatitis (affected is defined by physical examination findings: erythema, edema, scaling, lichenification, excoriation, with the excoriation serving as the physical examination correlate of pruritus) at Screening and Baseline.

   a. Subjects' BSA can include face and body OR body alone BUT NOT face alone.
7. An Investigator Global Assessment (IGA) score of 2-3 at Screening and Baseline.
8. Willing and able to complete once-daily eDiary entries within a consistent timeframe for the duration of the study and have ≥80% eDiary compliance rate during the washout period.
9. Judged to be in good health in the investigator's opinion.,

Exclusion Criteria:

1. Clearly defined etiology for pruritus other than atopic dermatitis. These include but are not limited to urticaria, psoriasis or other non-atopic dermatologic conditions, hepatic or renal disease, psychogenic pruritus, drug reaction, untreated hyperthyroidism, parasite presence and presence of acute infection either systemically or in the AD lesions.
2. Presence of any acute condition which may risk inducing an atopic dermatitis flare during the course of the study, such as impetigo or active herpes simplex infection.
3. Treatment with systemic corticosteroids within 4 weeks prior to randomization.
4. Treatment with Class III or higher potency topical corticosteroids or any topical anti-pruritic therapies (other than stable doses of low- or mid-potency topical corticosteroids or bland emollients) within 4 weeks prior to randomization.
5. Treatment with systemic therapies with recognized anti-pruritic (e.g. tricyclic antidepressants, sedatives, tranquilizers, gabapentin, marijuana or other cannabinoids, opioid receptor agonists/antagonists) or pruritic (e.g. opioids, angiotensin-converting enzyme inhibitors, cocaine,,antimalarials) properties within 4 weeks prior to randomization.

   a. Stable doses of H1 antihistamines will be permitted. Subjects must be willing to continue these at the same doses and frequencies throughout the study inclusive of the follow-up period.
6. Any clinically significant changes in type, dose, or frequency of bland emollients, low- or mid-potency corticosteroids, and/or oral H1 antihistamines throughout the study from screening to follow-up.
7. Treatment with systemic immunosuppressive/ immunomodulatory therapies within 4 weeks prior to randomization (including but not limited to phosphodiesterase-4 inhibitors, cyclosporine, mycophenolate-mofetil, methotrexate, azathioprine, interferon-gamma, or phototherapy).
8. Treatment with biologic therapies within 12 weeks or 5 half-lives prior to randomization, whichever is longer.
9. Use of an indoor tanning facility within 4 weeks prior to randomization.
10. Treatment with any investigational therapy within 4 weeks prior to randomization.
11. Allergen immunotherapy within 6 months prior to randomization.
12. Prior use of AO+ Mist.
13. History of malignancy within 5 years prior to randomization, with the exception of completely treated and non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin.
14. History of a major psychiatric condition (including major depressive disorder, bipolar disorder, or schizophrenia), suicidal ideation, or suicide attempt.
15. Known active hepatitis infection.
16. Known history of human immunodeficiency virus (HIV) infection.
17. Presence of any medical condition or disability that, in the investigator's opinion, could interfere with the assessment of safety or efficacy in this trial or compromise the safety of the subject.
18. Currently pregnant or breastfeeding, or male subject with a pregnant or breastfeeding partner.
19. Females of childbearing potential who are unable or unwilling to practice highly effective contraception (pregnancy prevention); fertile males who are unable or unwilling to use condoms with female partners of childbearing potential.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kim, PhD, Study Director — AOBiome LLC
Locations (56):
- United States (56):
  - Cahaba Dermatology, Birmingham, Alabama
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Cognitive Clinical Trials, Scottsdale, Arizona
  - Dermatology Trial Associates, Bryant, Arkansas
  - Applied Research Center of Arkansas, Inc, Little Rock, Arkansas
  - Core Healthcare Group, Cerritos, California
  - Encino Research Center, Encino, California
  - Center for Dermatology, INC, Fremont, California
  - Antelope Valley Clinical Trials, Lancaster, California
  - Long Beach Clinical Trials Services, Long Beach, California
  - L.A. Universal Research Center Inc, Los Angeles, California
  - Providence Clinical Research, North Hollywood, California
  - Syrentis Clinical Research, Santa Ana, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Tampa Bay Medical Research, Clearwater, Florida
  - Palm Beach Dermatology Group, Delray Beach, Florida
  - South Coast Research Center, Inc, Miami, Florida
  - D&H National Research Center, Miami, Florida
  - Meridian International Research, Miami Gardens, Florida
  - NAPA Research, Pompano Beach, Florida
  - Clinical Research Trials of Florida, Inc, Tampa, Florida
  - Moore Clinical Research, Tampa, Florida
  - Medical Dermatology Associates of Chicago, Chicago, Illinois
  - Clinical Investigation Specialists, Libertyville, Illinois
  - Sneeze Wheeze & Itch Associates, LLC, Normal, Illinois
  - Epiphany Dermatology, Overland Park, Kansas
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - Continental Clinical Solutions, Towson, Maryland
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - Clarkston Dermatology, Clarkston, Michigan
  - Onyx Clinical Reserach, Flint, Michigan
  - mediSearch Clinical Trials, Saint Joseph, Missouri
  - Thomas Dermatology, Henderson, Nevada
  - JDR Dermatology Research, LLC, Las Vegas, Nevada
  - ActivMed Practices & Research, Portsmouth, New Hampshire
  - The Dermatology Group, P. C., Verona, New Jersey
  - Drug Trials Brooklyn, Brooklyn, New York
  - Drug Trials America, Hartsdale, New York
  - Saddick Research Group, New York, New York
  - Dermatology Consulting Services, LLC, High Point, North Carolina
  - Wake Research, Raleigh, North Carolina
  - Clinical Research Solutions, Cleveland, Ohio
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Velocity Clinical Research, Medford, Oregon
  - Dermdox Centers for Dematology, Sugarloaf, Pennsylvania
  - Peak Research LLC, Upper Saint Clair, Pennsylvania
  - Greater Providence Clinical Research, Cranston, Rhode Island
  - AAPRI Research, Warwick, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Dermatology & Laser Center of Charleston, Charleston, South Carolina
  - Peak Research LLC, Fort Mill, South Carolina
  - Clinical Research Solutions, Milan, Tennessee
  - ACRC Trials, Plano, Texas
  - Aspen Dermatology, Orem, Utah
  - Advance Clinical Research, Salt Lake City, Utah
  - Dominion Medical Associates, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silverberg JI, Lio PA, Simpson EL, Li C, Brownell DR, Gryllos I, Ng-Cashin J, Krueger T, Swaidan VR, Bliss RL, Kim HD. Efficacy and safety of topically applied therapeutic ammonia oxidising bacteria in adults with mild-to-moderate atopic dermatitis and moderate-to-severe pruritus: a randomised, double-blind, placebo-controlled, dose-ranging, phase 2b trial. EClinicalMedicine. 2023 May 16;60:102002. doi: 10.1016/j.eclinm.2023.102002. eCollection 2023 Jun. PMID 37396805

RESULTS

PARTICIPANT FLOW:
Groups:
- B244 O.D. 5.0: B244 suspension (1x10E10 cells/ml) in 30ml/bottle
  Subjects will apply a total of 10 pumps of IP per application to all affected areas twice-a-day
  B244: B244 suspension
- B244 O.D. 20.0: B244 suspension (4x10E10 cells/ml) in 30ml/bottle
  Subjects will apply a total of 10 pumps of IP per application to all affected areas twice-a-day
  B244: B244 suspension
- Vehicle: Vehicle, 30ml/bottle
  Subjects will apply a total of 10 pumps of IP per application to all affected areas twice-a-day
  Vehicle: Vehicle suspension
Period: Overall Study
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Started | 180 | 180 | 187
Treated | 180 | 180 | 186
Completed | 161 | 155 | 166
Not Completed | 19 | 25 | 21
Not completed — Lost to Follow-up | 3 | 10 | 4
Not completed — Withdrawal by Subject | 8 | 6 | 9
Not completed — Physician Decision | 0 | 2 | 3
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Significant Non-Compliance | 2 | 4 | 4
Not completed — Significant Clinical Event | 0 | 1 | 0
Not completed — Other Reason | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Population includes patients from the Modified Intent-to-Treat (mITT) population, including all randomized participants who applied at least 1 dose of study medication and had at least one post-baseline evaluation on-site visit. Baseline measures collected include all measures that were collected under the study protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle | Total
Number analyzed (Participants) | 172 | 172 | 177 | 521
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (12.93) | 42.1 (13.49) | 42.1 (13.15) | 42.1 (13.17)
Age, Customized [Count of Participants; unit: Participants]
  18 to 40 years | 78 | 80 | 74 | 232
  41 to 54 years | 57 | 52 | 64 | 173
  55 to 65 years | 37 | 40 | 39 | 116
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 111 | 122 | 351
  Male | 54 | 61 | 55 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 87 | 88 | 85 | 260
  Not Hispanic or Latino | 85 | 84 | 92 | 261
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 19 | 18 | 21 | 58
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 36 | 41 | 39 | 116
  White | 113 | 111 | 114 | 338
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 2 | 8
Height [Mean (Standard Deviation); unit: centimeters] | 166.100 (9.706) | 165.608 (9.923) | 166.102 (8.836) | 165.938 (9.479)
Weight [Mean (Standard Deviation); unit: kilograms] | 84.144 (22.104) | 81.351 (19.603) | 81.908 (20.653) | 82.462 (20.805)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/meters^2] | 30.576 (8.112) | 29.610 (6.577) | 29.729 (7.403) | 29.969 (7.389)
Body Surface Area (BSA) [Count of Participants; unit: Participants]
  10-20% | 108 | 113 | 118 | 339
  >20-30% | 53 | 52 | 52 | 157
  >30-40% | 11 | 7 | 7 | 25
Body Surface Area (BSA) [Mean (Standard Deviation); unit: percentage of body surface] | 18.82 (7.247) | 18.02 (6.069) | 18.08 (6.600) | 18.30 (6.653)
Smoking Status [Count of Participants; unit: Participants]
  Yes | 30 | 28 | 29 | 87
  No | 142 | 144 | 148 | 434
Rescue Medication [Count of Participants; unit: Participants]
  Yes | 30 | 27 | 33 | 90
  No | 142 | 145 | 144 | 431
Rescue Medication Days [Mean (Standard Deviation); unit: days] — Population: The population analyzed in this row represents only the participants who used a rescue medication.
  days
    number analyzed (Participants) | 30 | 27 | 33 | 90
    (all) | 1.4 (0.72) | 1.3 (0.78) | 1.7 (1.85) | 1.5 (1.26)
Worst Itch Numeric Rating Scale (WI-NRS) [Mean (Standard Deviation); unit: score on a scale] — The Itch Numeric Rating Scale (I-NRS) is a validated, self-reported instrument for measurement of itch intensity. It uses a 24-hour recall period and asks subjects to rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicate greater itch intensity. Worst itch intensity (WI-NRS) during a 24-hour recall period will be captured. The question for WI-NRS would be, "Please rate the itching severity due to your atopic dermatitis by circling the number that best describes your worst level of itching in the past 24 hours."
  score on a scale | 8.21 (0.913) | 8.26 (1.004) | 8.26 (1.094) | 8.24 (1.006)
Average Itch Numeric Rating Scale (AI-NRS) [Mean (Standard Deviation); unit: score on a scale] — The Itch Numeric Rating Scale (I-NRS) is a validated, self-reported instrument for measurement of itch intensity. It uses a 24-hour recall period and asks subjects to rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicate greater itch intensity. Average itch intensity (AI-NRS) during a 24-hour recall period will be captured. The question for AI-NRS would be, "Please rate the itching severity due to your atopic dermatitis by circling the number that best describes your average level of itching in the past 24 hours."
  score on a scale | 7.53 (1.062) | 7.42 (1.344) | 7.39 (1.374) | 7.45 (1.268)
5-D Pruritus Scale Total Score [Mean (Standard Deviation); unit: score on a scale] — The 5-D Pruritus Scale is a validated, multi-dimensional measure of itching that assesses the five domains of degree, duration, direction, disability, and distribution. The domains are scored separately and then summed together to obtain a total 5-D score, ranging from 5 (no pruritus) to 25 (most severe pruritus).
  score on a scale | 17.0 (2.59) | 16.6 (2.86) | 17.0 (2.89) | 16.9 (2.79)
Eczema Area Severity Index (EASI) [Count of Participants; unit: Participants] — Eczema Area Severity Index (EASI) is a validated tool used to measure the severity and extent of atopic dermatitis where clinical investigators assess the presence and severity of erythema, edema/papulation, excoriation, and lichenification and area of involvement across head and neck, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks). The EASI score can range from 0.0 to 72.0 with increments of 0.1 and higher scores representing a greater severity of atopic dermatitis.
  Participants
    <=10 | 125 | 116 | 122 | 363
    >10 | 47 | 56 | 55 | 158
Eczema Area Severity Index (EASI) Total Score [Mean (Standard Deviation); unit: score on a scale] — Eczema Area Severity Index (EASI) is a validated tool used to measure the severity and extent of atopic dermatitis where clinical investigators assess the presence and severity of erythema, edema/papulation, excoriation, and lichenification and area of involvement across head and neck, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks). The EASI score can range from 0.0 to 72.0 with increments of 0.1 and higher scores representing a greater severity of atopic dermatitis.
  score on a scale | 9.23 (5.463) | 8.98 (4.321) | 8.92 (4.560) | 9.04 (4.797)
Investigator's Global Assessment (IGA) [Count of Participants; unit: Participants] — Investigator's Global Assessment (IGA) was used to assess the overall diseases severity on a scale of 0 to 4 (0=clear, 1=almost clear, 2=mild disease, 3=moderate disease, and 4=severe disease).
  Participants
    Mild | 53 | 53 | 48 | 154
    Moderate | 117 | 119 | 129 | 365
    Severe | 2 | 0 | 0 | 2
Investigator's Global Assessment (IGA) [Mean (Standard Deviation); unit: score on a scale] — Investigator's Global Assessment (IGA) was used to assess the overall diseases severity on a scale of 0 to 4 (0=clear, 1=almost clear, 2=mild disease, 3=moderate disease, and 4=severe disease).
  score on a scale | 2.7 (0.48) | 2.7 (0.46) | 2.7 (0.45) | 2.7 (0.46)
Patient Oriented Eczema Measure (POEM) Total Score [Mean (Standard Deviation); unit: score on a scale] — The Patient Oriented Eczema Measure (POEM) is a tool developed by the University of Nottingham, United Kingdom, for monitoring atopic dermatitis severity. The subject will complete the questionnaire at each of the assessment timepoints as outlined. Each of the 7 questions in the POEM questionnaire carries equal weight and is scored from 0 to 4: No days = 0. 1 to 2 days = 1. 3 to 4 days = 2. 5 to 6 days = 3. Every day = 4. Scores are then added to yield a total score of 0 to 28; higher scores mean the greater the severity of atopic dermatitis.
  score on a scale | 16.6 (5.03) | 15.7 (4.88) | 16.1 (5.49) | 16.1 (5.14)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Worst Itch Numeric Rating Scale (WI-NRS)
Description: The Itch Numeric Rating Scale (I-NRS) is a validated, self-reported instrument for measurement of itch intensity. It uses a 24-hour recall period and asks subjects to rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicate greater itch intensity. Worst itch intensity (WI-NRS) during a 24-hour recall period will be captured. The question for WI-NRS would be, "Please rate the itching severity due to your atopic dermatitis by circling the number that best describes your worst level of itching in the past 24 hours."
Time Frame: Baseline to Day 28
Population: Subjects from the Modified Intent to Treat (mITT) population (all randomized participants who applied at least 1 dose of study medication and had at least one post-baseline evaluation on-site visit. Subjects were grouped as randomized) that remained in the study at Day 28
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 166 | 165 | 174
score on a scale | -2.8 (0.184) | -2.8 (0.184) | -2.1 (0.180)
Statistical Analysis 1: Comparison: B244 O.D. 5.0 vs Vehicle; Approximately 576 subjects may be enrolled to account for 16.7% drop out rate prior to completing the study. A total of 160 evaluable subjects per group are required to achieve at least 80% power to detect a difference of 0.65 in mean WI-NRS change from Baseline to Week 4 between one of two active doses of B244 and vehicle control when assuming a standard deviation of 2.5 and applying a Dunnett Testing Method at a one-sided familywise error rate of 0.10; Test type: Superiority — The ANCOVA model for primary endpoint change from Baseline to Week 4 in average WI-NRS will have treatment group and Baseline weekly average WI-NRS as explanatory variables. Hypothesis will be tested using a Dunnett Testing Method, applying pairwise comparisons of each group to vehicle using a one-sided familywise error rate of 0.10. Treatment effect will be estimated as least squares means using vehicle as reference and adjusted using Dunnett Testing Method and presented with one-sided 90% CI; p = 0.0148, ANCOVA
Statistical Analysis 2: Comparison: B244 O.D. 20.0 vs Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0143, ANCOVA

2. Secondary Outcome: Proportion of Patients With ≥4 Point Improvement in Worst Itch Numeric Rating Scale (WI-NRS)
Description: as for outcome 1
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 166 | 165 | 174
Participants | 51 | 51 | 38

3. Secondary Outcome: Proportion of Subjects With Any Improvement in Worst Itch Numeric Rating Scale (WI-NRS)
Description: as for outcome 1
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 166 | 165 | 174
Participants | 120 | 115 | 105
Statistical Analysis 1: Comparison: B244 O.D. 5.0 vs Vehicle; The frequency and rate of WI-NRS and AI-NRS responders will be reported and compared between treatment groups using a logistic regression model. Generalized estimating equations to account for repeated measures and within-subject variability may also be applied; Test type: Superiority; p = 0.0205, Regression, Logistic

4. Secondary Outcome: Mean Change in Average Itch Numeric Rating Scale (AI-NRS)
Description: The Itch Numeric Rating Scale (I-NRS) is a validated, self-reported instrument for measurement of itch intensity. It uses a 24-hour recall period and asks subjects to rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable). Higher scores indicate greater itch intensity. Average itch intensity (AI-NRS) during a 24-hour recall period will be captured. The question for AI-NRS would be, "Please rate the itching severity due to your atopic dermatitis by circling the number that best describes your average level of itching in the past 24 hours."
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 165 | 164 | 172
score on a scale | -2.7 (.132) | -2.7 (.132) | -2.1 (.164)
Statistical Analysis 1: Comparison: B244 O.D. 5.0 vs Vehicle; The difference in treatment groups in change from Baseline values at post-baseline visits will be analyzed using a mixed model with repeated measures; Test type: Superiority; p = 0.0044, Mixed Models Analysis
Statistical Analysis 2: Comparison: B244 O.D. 20.0 vs Vehicle; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0077, Mixed Models Analysis

5. Secondary Outcome: Proportion of Subjects With ≥4 Point Improvement in Average Itch Numeric Rating Scale (AI-NRS)
Description: as for outcome 4
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 165 | 164 | 172
Participants | 54 | 53 | 39
Statistical Analysis 1: Comparison: B244 O.D. 5.0 vs Vehicle; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0400, Regression, Logistic
Statistical Analysis 2: Comparison: B244 O.D. 20.0 vs Vehicle; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0486, Regression, Logistic

6. Secondary Outcome: Proportion of Subjects With Any Improvement in Average Itch Numeric Rating Scale (AI-NRS)
Description: as for outcome 4
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 165 | 164 | 172
Participants | 118 | 112 | 110

7. Secondary Outcome: Mean Change in Worst Itch Numeric Rating Scale (WI-NRS)
Description: as for outcome 1
Time Frame: Baseline to Day 14
Population: Subjects from the Modified Intent to Treat (mITT) population (all randomized participants who applied at least 1 dose of study medication and had at least one post-baseline evaluation on-site visit. Subjects were grouped as randomized) that remained in the study at Day 14
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 170 | 172 | 174
score on a scale | -2.0 (.138) | -2.0 (.137) | -1.5 (.170)
Statistical Analysis 1: Comparison: B244 O.D. 5.0 vs Vehicle; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0246, Mixed Models Analysis
Statistical Analysis 2: Comparison: B244 O.D. 20.0 vs Vehicle; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0366, Mixed Models Analysis

8. Secondary Outcome: Proportion of Subjects With ≥4 Point Improvement in Worst Itch Numeric Rating Scale (WI-NRS)
Description: as for outcome 1
Time Frame: Baseline to Day 14
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 170 | 172 | 174
Participants | 34 | 30 | 21
Statistical Analysis 1: Comparison: B244 O.D. 5.0 vs Vehicle; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0467, Regression, Logistic

9. Secondary Outcome: Mean Change in Patient Oriented Eczema Measure (POEM)
Description: The Patient Oriented Eczema Measure (POEM) is a tool developed by the University of Nottingham, United Kingdom, for monitoring atopic dermatitis severity. The subject will complete the questionnaire at each of the assessment timepoints as outlined. Each of the 7 questions in the POEM questionnaire carries equal weight and is scored from 0 to 4: No days = 0. 1 to 2 days = 1. 3 to 4 days = 2. 5 to 6 days = 3. Every day = 4. Scores are then added to yield a total score of 0 to 28; higher scores mean the greater the severity of atopic dermatitis.
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 166 | 164 | 171
score on a scale | -6.4 (.342) | -6.0 (.343) | -5.2 (.394)
Statistical Analysis 1: Comparison: B244 O.D. 5.0 vs Vehicle; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0293, Mixed Models Analysis

10. Secondary Outcome: Mean Change in 5-D Pruritus Scale
Description: The 5-D Pruritus Scale is a validated, multi-dimensional measure of itching that assesses the five domains of degree (score 1-5: 1=not present, 2=mild, 3=moderate, 4=severe, 5=unbearable), duration (score 1-5: 1=less than 6hrs/day, 2=6-12hrs/day, 3=12-18hrs/day, 4=18-23hrs/day, 5=all day), direction (score 1-5: 1=completely resolved, 2=much better/still present, 3=little bit better/still present, 4=unchanged, 5=getting worse), disability (score 1-5: 1=never affects activity, 2=rarely affects activity, 3=occasionally affects activity, 4=frequently affects activity, 5=always affects activity; highest activity score is taken), and distribution (check boxes of affected body parts; 0-2 body parts=score of 1, 3-5=score of 2, 6-10=score of 3, 11-13=score of 4, 14-16=score of 5).
  The domains are scored separately and then summed together to obtain a total 5-D score, ranging from 5 (no pruritus) to 25 (most severe pruritus). Subjects rate their symptoms over the preceding 2-week period.
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 166 | 164 | 171
score on a scale | -5.2 (.228) | -5.2 (.229) | -4.2 (.262)
Statistical Analysis 1: Comparison: B244 O.D. 5.0 vs Vehicle; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0045, Mixed Models Analysis
Statistical Analysis 2: Comparison: B244 O.D. 20.0 vs Vehicle; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0043, Mixed Models Analysis

11. Other Pre Specified Outcome: Mean Change in Investigator's Global Assessment (IGA)
Description: Investigator's Global Assessment (IGA) was used to assess the overall diseases severity on a scale of 0 to 4 (0=clear, 1=almost clear, 2=mild disease, 3=moderate disease, and 4=severe disease).
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 166 | 164 | 171
score on a scale | -0.8 (.056) | -0.8 (.056) | -0.5 (.064)
Statistical Analysis 1: Comparison: B244 O.D. 5.0 vs Vehicle; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0026, Mixed Models Analysis
Statistical Analysis 2: Comparison: B244 O.D. 20.0 vs Vehicle; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0005, Mixed Models Analysis

12. Other Pre Specified Outcome: Mean Change in Eczema Area Severity Index (EASI)
Description: Eczema Area Severity Index (EASI) is a validated tool used to measure the severity and extent of atopic dermatitis where clinical investigators assess the presence and severity of erythema, edema/papulation, excoriation, and lichenification (score 0-3: none=0, mild=1, moderate=2, severe=3, half-points allowed) and area of involvement (score 0-6: 0=0% involvement, 1=1-9% involvement, 2=10-29% involvement, 3=30-49% involvement, 4=50-69% involvement, 5=70-89% involvement, 6=90-100% involvement) across head and neck, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks). The EASI score can range from 0.0 to 72.0 with increments of 0.1 and higher scores representing a greater severity of atopic dermatitis.
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 166 | 164 | 171
score on a scale | -3.9 (.249) | -4.0 (.250) | -3.1 (.289)
Statistical Analysis 1: Comparison: B244 O.D. 5.0 vs Vehicle; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0348, Mixed Models Analysis
Statistical Analysis 2: Comparison: B244 O.D. 20.0 vs Vehicle; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0173, Mixed Models Analysis

13. Other Pre Specified Outcome: Proportion of Subjects With Investigator's Global Assessment (IGA) of Clear or Almost Clear and ≥2 Point Improvement
Description: as for outcome 11
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 166 | 164 | 171
Participants | 36 | 43 | 21
Statistical Analysis 1: Comparison: B244 O.D. 5.0 vs Vehicle; Responder rates for IGA and EASI will be summarized using descriptive statistics and analyzed using a logistic regression model at each respective timepoints; Test type: Superiority; p = 0.0228, Regression, Logistic
Statistical Analysis 2: Comparison: B244 O.D. 20.0 vs Vehicle; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0015, Regression, Logistic

14. Other Pre Specified Outcome: Proportion of Subjects With Investigator's Global Assessment (IGA) of Clear or Almost Clear at Week 4
Description: as for outcome 11
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 166 | 164 | 171
Participants | 46 | 62 | 34
Statistical Analysis 1: Comparison: B244 O.D. 20.0 vs Vehicle; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0003, Regression, Logistic

15. Other Pre Specified Outcome: Proportion of Subjects With Any Improvement in Investigator's Global Assessment (IGA) From Baseline to Week 4
Description: as for outcome 11
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 166 | 164 | 171
Participants | 81 | 91 | 73
Statistical Analysis 1: Comparison: B244 O.D. 20.0 vs Vehicle; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0195, Regression, Logistic

16. Other Pre Specified Outcome: Proportion of Subjects With ≥50% Improvement in Eczema Area Severity Index (EASI-50)
Description: as for outcome 12
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 166 | 164 | 171
Participants | 74 | 76 | 60
Statistical Analysis 1: Comparison: B244 O.D. 20.0 vs Vehicle; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0365, Regression, Logistic

17. Other Pre Specified Outcome: Proportion of Subjects With ≥75% Improvement in Eczema Area Severity Index (EASI-75)
Description: as for outcome 12
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 166 | 164 | 171
Participants | 46 | 48 | 27
Statistical Analysis 1: Comparison: B244 O.D. 5.0 vs Vehicle; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0086, Regression, Logistic
Statistical Analysis 2: Comparison: B244 O.D. 20.0 vs Vehicle; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0035, Regression, Logistic

18. Other Pre Specified Outcome: Proportion of Subjects With ≥90% Improvement in Eczema Area Severity Index (EASI-90)
Description: as for outcome 12
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
Number analyzed (Participants) | 166 | 164 | 171
Participants | 25 | 30 | 10
Statistical Analysis 1: Comparison: B244 O.D. 5.0 vs Vehicle; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0074, Regression, Logistic
Statistical Analysis 2: Comparison: B244 O.D. 20.0 vs Vehicle; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.0008, Regression, Logistic

ADVERSE EVENTS:
Time Frame: Screening visit to Week 8.
Description: All adverse events (AEs) occurring after signing of the ICF through study completion/early termination were to be reported. All AEs were to be recorded irrespective of whether they were considered drug related. AEs were to be evaluated by the Investigator at each visit for duration, intensity, and whether the event could have been associated with the IP or other causes. AEs believed to be possibly related to IP must have been followed until their resolution.
Arm/Group | B244 O.D. 5.0 | B244 O.D. 20.0 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/180 | 0/186
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/180 | 0/186
Other Adverse Events (participants affected / at risk) | 33/180 | 29/180 | 17/186
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B244 O.D. 5.0 (N=180) | B244 O.D. 20.0 (N=180) | Vehicle (N=186)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1 | 0
Application site dryness (General disorders) | 0 | 0 | 1
Application site erythema (General disorders) | 2 | 0 | 0
Application site pain (General disorders) | 1 | 1 | 2
Application site pruritus (General disorders) | 3 | 0 | 0
Application site rash (General disorders) | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Vaccination site discomfort (General disorders) | 3 | 0 | 1
Food allergy (Immune system disorders) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 3 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 2
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 6 | 4 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Cataract operation (Surgical and medical procedures) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall have 60 days to review the papers. Sponsor shall have the right to require Institution/Principal Investigator, as applicable, to remove specifically identified confidential information and/or delay the proposed publication or presentation for an additional 90 days to enable Sponsor to seek patent protections.

DOCUMENTS (2):
  • Study Protocol (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT04490109/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT04490109/SAP_002.pdf